CLINICAL TRIAL: NCT04863794
Title: A Non-Randomized, Open-Label, Adaptive, Single Center, Positron Emission Tomography (Pet) Study To Assess Distribution Of RO7248824 In The Central Nervous System Following Single Intrathecal Doses Of [89zr] Labeled RO7248824 In Healthy Male Participants
Brief Title: A Study To Assess Distribution Of RO7248824 In The Central Nervous System Following Single Intrathecal Doses Of [89zr] Labeled RO7248824 In Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP41660
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RO7248824 (Experimental): In Part 1 of the study RO7248824 and [89Zr]-labeled RO7248824 will be administered as a single bolus IT injection following a standard IT Administration procedure. In Part 2 of the study, it is planned to test up to 3 additional IT procedures. This part is tentative with regard to its conduct and the number of procedures that may be tested.
  Interventions: Drug: RO7248824

INTERVENTIONS:
Drug: RO7248824 — A single dose of 10 mg RO7248824 will be used for this PET study in healthy participants.

SUMMARY:
The aim of Study BP41660 is to quantify the amount and concentration of [89Zr]DFO-RO7248824 in the brain with positron emission tomography (PET) following a single sub-pharmacological dose of RO7248824 and [89Zr]DFO-RO7248824 administered via IT injection to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent

1. Able and willing to provide written informed consent and to comply with the study protocol according to ICH and local regulations

   Age
2. Aged from 25 to to 55 years at the time of dosing

   Type of Participants and Disease Characteristics
3. Overtly healthy (defined by absence of evidence of any active or chronic disease) as determined by medical evaluation including:

   * A detailed medical and surgical history
   * A complete physical and neurological examination
   * Vital signs
   * 12-lead ECG
   * Hematology
   * Coagulation
   * Blood chemistry
   * Serology and urinalysis
4. Fluent in the language of the Investigator and study staff, and able to communicate with the study staff

   Weight
5. Body mass index (BMI) of ≥ 18 to ≤ 30 kg/m2 at screening

   Sex
6. Male participants only who, for 3 months after the dosing of RO7248824, agree to:

   * Remain abstinent (refrain from heterosexual intercourse) or use contraceptive barrier measures such as a condom, with a female partner of childbearing potential, or pregnant female partner, to avoid exposing the embryo
   * Refrain from donating sperm

Exclusion Criteria:

Medical Conditions

1. Any condition or disease detected during the medical interview/physical examination that would render the participant unsuitable for the study, place the participant at undue risk or interfere with the ability of the participant to complete the study, as determined by the Investigator
2. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data
3. History or presence of clinically significant cardiovascular disease in the opinion of the Investigator
4. History or presence of an abnormal ECG that is clinically significant in the Investigator's opinion
5. Uncontrolled arrhythmias or history of clinically significant arrhythmias
6. Confirmed abnormal blood pressure
7. Abnormal pulse rate
8. Abnormalities in brain and
9. Evidence or history of clinically significant back pain, back pathology and/or back injury
10. Evidence or history of significant active bleeding or coagulation disorder
11. Allergy to lidocaine (Xylocaine) or its derivatives
12. Medical or surgical conditions for which LP or associated procedures is contraindicated
13. Alanine transaminase (ALT) and bilirubin > 1.5 x upper limit of normal (ULN)
14. Current or chronic history of liver disease, or known hepatic or biliary abnormalities
15. History of convulsions or history of loss of consciousness
16. Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates the participation in the study
17. Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first study drug administration
18. Clinically significant abnormalities in laboratory test results

    Prior/Concomitant Therapy
19. Used or intends to use any prohibited medications
20. Likely to need concomitant medication during the study period

    Prior/Concurrent Clinical Study Experience
21. Participating in an investigational drug or device study within 60 days prior to screening, as calculated from the day of follow-up from the previous study, or more than 4 participations in an investigational drug or device study within a year prior to dosing
22. Previously (within the past 12 months from dosing) included in medical research and/or a medical protocol involving PET or radiological investigations, or other exposure to ionizing radiation, which combined with this study would result in an effective dose of 10 mSv or more

    Diagnostic Assessments
23. Positive test for drugs of abuse or alcohol
24. Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment)
25. Evidence of HIV infection and/or positive human HIV antibodies

    Other Exclusions
26. Any suspicion or history of alcohol abuse and/or suspicion of regular consumption of drug of abuse or previous history of or treatment for a dependence disorder
27. Regularly smoking more than 5 cigarettes daily or equivalent and unable or unwilling not to smoke or not to use other nicotine containing products during the in-house period
28. Donated over 500 mL of blood or blood products or had significant blood loss within 3 months prior to screening
29. Under judicial supervision, guardianship or curatorship
30. Not able to undergo PET, CT, or MRI scans
31. Previous lumbar surgery that is likely, in the opinion of the Investigator or surgical team, to make IT injection unduly difficult or hazardous
32. Scoliosis or spinal deformity preventing IT injection

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Quantification of [89Zr]DFO-RO7248824 distribution within the central nervous system (CNS) | Baseline up to 6 weeks

SECONDARY OUTCOMES:
Percentage of participants with adverse events (AEs) | Baseline up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Pra International Group B.V, Groningen, Netherlands